CLINICAL TRIAL: NCT01604824
Title: A Phase 2 Pilot Study With a Randomized Double-Blind Treatment Phase to Evaluate the Pharmacodynamics and Safety of Alirocumab in Patients With Autosomal Dominant Hypercholesterolemia and Gain-of-Function Mutations in 1 or Both Alleles of the PCSK9 Gene or Loss-of-Function Mutations in 1 or More Alleles of the Loss-of-Function Mutations B Gene
Brief Title: A Study of Alirocumab in Participants With Autosomal Dominant Hypercholesterolemia (ADH) and Gain-of-Function Mutations (GOFm) of the Proprotein Convertase Subtilisin Kexin 9 (PCSK9) Gene or Loss-of-Function Mutations (LOFm) of the Apolipoprotein (Apo) B Gene
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R727-CL-1018
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Results first posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (4):
- GOFm PCSK9 (Cohort 1): Alirocumab From Day 1 (Experimental): Participants with gain-of-function mutation (GOFm) in proprotein convertase subtilisin/kexin type 9 (PCSK9) gene (Cohort 1): Alirocumab 150 mg subcutaneous (SC) injection at Week 0 (Day 1), Week 2 (Day 15), Week 4, 6 and 10 (matching placebo at Week 8, 12 and 14) during the double-blind period (Group A). Afterwards, participants have the possibility to continue in an open-label extension period with 150 mg alirocumab SC twice per week (Q2W) for an additional 3 years.
  Interventions: Drug: Alirocumab; Drug: Placebo
- GOFm PCSK9 (Cohort 1): Alirocumab From Day 15 (Experimental): Participants with gain-of-function mutation (GOFm) in proprotein convertase subtilisin/kexin type 9 (PCSK9) gene (Cohort 1): Alirocumab 150 mg subcutaneous (SC) injection at Week 2 (Day 15), Week 4, 6, 8 and 12 ([matching placebo at Week 0 (Day 1), 10 and 14]) during the double-blind period (Group B). Afterwards, participants have the possibility to continue in an open-label extension period with 150 mg alirocumab SC twice per week (Q2W) for an additional 3 years.
  Interventions: Drug: Alirocumab; Drug: Placebo
- GOFm PCSK9 or LOFm ApoB (Cohort 2): Alirocumab from Day 1 (Experimental): Participants with gain-of-function mutation (GOFm) in the proprotein convertase subtilisin/kexin type 9 (PCSK9) gene or loss-of-function mutation (LOFm) in the apolipoprotein (Apo) B gene (Cohort 2): Alirocumab 150 mg subcutaneous (SC) injection at Week 0 (Day 1), Week 2 (Day 15), Week 4, 6 and 10 (matching placebo at Week 8, 12 and 14) during the double-blind period (Group C). Afterwards, participants have the possibility to continue in an open-label extension period with 150 mg alirocumab SC twice per week (Q2W) for an additional 3 years.
  Interventions: Drug: Alirocumab; Drug: Placebo
- GOFm PCSK9 or LOFm ApoB (Cohort 2): Alirocumab from Day 15 (Experimental): Participants with gain-of-function mutation (GOFm) in proprotein convertase subtilisin/kexin type 9 (PCSK9) gene or loss-of-function mutation (LOFm) in apolipoprotein (Apo) B gene (Cohort 2): Alirocumab 150 mg subcutaneous (SC) injection at Week 2 (Day 15), Week 4, 6, 8 and 12 ([matching placebo at Week 0 (Day 1), 10 and 14]) during the double-blind period (Group D). Afterwards, participants have the possibility to continue in an open-label extension period with 150 mg alirocumab SC twice per week (Q2W) for an additional 3 years.
  Interventions: Drug: Alirocumab; Drug: Placebo

INTERVENTIONS:
Drug: Alirocumab — SC injection in the abdomen
  Other Names: Praluent®; REGN727; SAR236553
Drug: Placebo — SC injection in the abdomen

SUMMARY:
The primary objective of the study is to assess the pharmacodynamic (PD) effect of alirocumab on serum low density lipoprotein cholesterol (LDL-C) during 14 weeks of subcutaneous (SC) administered alirocumab in patients with autosomal dominant hypercholesterolemia (ADH) and gain-of-function mutation (GOFm) in 1 or both alleles of the proprotein convertase subtilisin/kexin type 9 (PCSK9) gene or with loss-of-function mutation (LOFm) in 1 or more alleles of the apolipoprotein (ApoB) gene.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include, but are not limited to the following:

1. Between the ages of 18 and 70 years, inclusive
2. A history of molecularly confirmed PCSK9 GOFm for cohort 1 and a history of molecularly confirmed PCSK9 GOFm or ApoB LOFm
3. Plasma LDL-Cholesterol levels ≥70 mg/dL at the screening visit on a lipid-lowering therapy (LLT) regimen stable for at least 28 days

Exclusion Criteria:

Exclusion criteria include, but are not limited to the following:

1. Serum triglycerides >350 mg/dL at the screening visit
2. Known to be positive for human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus
3. Pregnant or breast-feeding women.
4. Sexually active man or woman of childbearing potential who is unwilling to practice adequate contraception during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-02-22 (Actual); Primary Completion 2014-06-02 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (4):
- Salt Lake City, Utah, United States
- France (3):
  - Lille, Cedex
  - Nantes, Cedex
  - Paris

REFERENCES:
- [Derived] Hopkins PN, Krempf M, Bruckert E, Donahue S, Yang F, Zhang Y, DiCioccio AT. Pharmacokinetic and pharmacodynamic assessment of alirocumab in patients with familial hypercholesterolemia associated with proprotein convertase subtilisin/kexin type 9 gain-of-function or apolipoprotein B loss-of-function mutations. J Clin Lipidol. 2019 Nov-Dec;13(6):970-978. doi: 10.1016/j.jacl.2019.10.007. Epub 2019 Oct 21. PMID 31767518
- [Derived] Hopkins PN, Defesche J, Fouchier SW, Bruckert E, Luc G, Cariou B, Sjouke B, Leren TP, Harada-Shiba M, Mabuchi H, Rabes JP, Carrie A, van Heyningen C, Carreau V, Farnier M, Teoh YP, Bourbon M, Kawashiri MA, Nohara A, Soran H, Marais AD, Tada H, Abifadel M, Boileau C, Chanu B, Katsuda S, Kishimoto I, Lambert G, Makino H, Miyamoto Y, Pichelin M, Yagi K, Yamagishi M, Zair Y, Mellis S, Yancopoulos GD, Stahl N, Mendoza J, Du Y, Hamon S, Krempf M, Swergold GD. Characterization of Autosomal Dominant Hypercholesterolemia Caused by PCSK9 Gain of Function Mutations and Its Specific Treatment With Alirocumab, a PCSK9 Monoclonal Antibody. Circ Cardiovasc Genet. 2015 Dec;8(6):823-31. doi: 10.1161/CIRCGENETICS.115.001129. Epub 2015 Sep 15. PMID 26374825

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 4 sites, 3 in France & 1 in the United States. Twenty-eight participants were screened between Feb 2012 & Apr 2013. A total of 23 participants were enrolled: 13 in cohort 1 & 10 in cohort 2. Recruitment for cohort 2 occurred after the un-blinding of cohort 1 & analyses of the double-blind study data for cohort 1.
Pre-assignment Details: Eligible participants entered a 2-wk, single-blind, placebo run-in period. Participants in cohort 1 were randomized in a 1:1 ratio (group A or B); Participants in cohort 2 were also randomized in a 1:1 ratio (group C or D).
Groups:
- PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A): Participants with a gain-of-function mutation (GOFm) in the PCSK9 gene (Cohort 1: Group A) received 150 mg alirocumab subcutaneously (SC) on days 1, 15, 29, 43, and 71 and matching placebo SC on days 57, 85, and 99 during the double-blind period. Participants who continued in an open-label extension period received 150 mg alirocumab SC twice per week (Q2W) for an additional 3 years.
- PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B): Participants with a GOFm in PCSK9 gene (Cohort 1: Group B) received 150 mg alirocumab SC on days 15, 29, 43, 57, and 85 and matching placebo SC on days 1, 71, and 99 during the double-blind period. Participants who continued in an open-label extension period received 150 mg alirocumab SC twice per week (Q2W) for an additional 3 years.
- PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C): Participants with a GOFm in the PCSK9 gene or a LOFm in the Apo B gene (Cohort 2: Group C) received 150 mg alirocumab SC on days 1, 15, 29, 43, and 71 and matching placebo SC on days 57, 85, and 99. Participants who continued in an open-label extension period received 150 mg alirocumab SC twice per week (Q2W) for an additional 3 years.
- PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2: Group D): Participants with a GOFm in PCSK9 gene or LOFm in Apo B gene (Cohort 2: Group D) received 150 mg alirocumab SC on days 15, 29, 43, 57, and 85 and matching placebo SC on days 1, 71, and 99 during the double-blind period. Participants who continued in an open-label extension period received 150 mg alirocumab SC twice per week (Q2W) for an additional 3 years.
- PCSK9 GOFm (Cohort 1: Group A and Group B): Participants with a GOFm in the PCSK9 gene (Cohort 1: Group A) received 150 mg alirocumab subcutaneously (SC) on days 1, 15, 29, 43, and 71 and matching placebo SC on days 57, 85, and 99 during the double-blind period. Participants with a GOFm in PCSK9 gene (Cohort 1: Group B) received 150 mg alirocumab SC on days 15, 29, 43, 57, and 85 and matching placebo SC on days 1, 71, and 99 during the double-blind period. Participants who continued in an open-label extension period received 150 mg alirocumab SC, Q2W for an additional 3 years.
- PCSK9 GOFm/ApoB LOFm (Cohort 2: Group C and Group D): Participants with a GOFm in the PCSK9 gene or a LOFm in the Apo B gene (Cohort 2: Group C) received 150 mg alirocumab SC on days 1, 15, 29, 43, and 71 and matching placebo SC on days 57, 85, and 99. Participants with a GOFm in PCSK9 gene or LOFm in Apo B gene (Cohort 2: Group D) received 150 mg alirocumab SC on days 15, 29, 43, 57, and 85 and matching placebo SC on days 1, 71, and 99 during the double-blind period. Participants who continued in an open-label extension period received 150 mg alirocumab SC twice per week (Q2W) for an additional 3 years.
Period: Double-blind (DB) Period
Arm/Group | PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) | PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B) | PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) | PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2: Group D) | PCSK9 GOFm (Cohort 1: Group A and Group B) | PCSK9 GOFm/ApoB LOFm (Cohort 2: Group C and Group D)
Started | 6 | 7 | 5 | 5 | 0 | 0
Completed DB Period (Day 99) | 6 | 7 | 5 | 5 | 0 | 0
Completed DB Follow-up (Day 155) | 6 | 7 | 5 | 5 | 0 | 0
Completed | 6 | 7 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-label Extension (OLE) Period
Arm/Group | PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) | PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B) | PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) | PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2: Group D) | PCSK9 GOFm (Cohort 1: Group A and Group B) | PCSK9 GOFm/ApoB LOFm (Cohort 2: Group C and Group D)
Started | 0 | 0 | 0 | 0 | 13 (Completed DB Period (Day 99)) | 10 (Completed DB follow-up (Day 155))
Started Open-label Extension Period | 0 | 0 | 0 | 0 | 11 (Two subjects chose not to enter OLE period) | 10
Completed Study | 0 | 0 | 0 | 0 | 10 | 10
Completed | 0 | 0 | 0 | 0 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Chose not to enter OLE Period | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Refused to come into office | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) | PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B) | PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) | PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2: Group D) | Total
Number analyzed (Participants) | 6 | 7 | 5 | 5 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (14.72) | 46.4 (13.24) | 45.6 (3.21) | 42.0 (10.84) | 44.2 (11.15)
Age, Customized [Number; unit: Participants]
  In utero | 0 | 0 | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0 | 0 | 0
  Adults (18-64 years) | 6 | 7 | 5 | 5 | 23
  From 65-84 years | 0 | 0 | 0 | 0 | 0
  85 years and over | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 2 | 15
  Male | 2 | 2 | 1 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 7 | 5 | 5 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  White | 5 | 6 | 5 | 5 | 21
  Black or African American | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other: Indian Ocean Islander | 0 | 1 | 0 | 0 | 1
  Other: Mauritius | 1 | 0 | 0 | 0 | 1
Measured Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Baseline value is defined as the last available value prior to the first dose of double-blind period (alirocumab or placebo).
  milligrams per deciliter (mg/dL) | 108.8 (33.84) | 144.3 (68.39) | 187.4 (98.12) | 151.0 (82.70) | 145.9 (72.82)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Baseline value is defined as the last available value prior to the first dose of double-blind period (alirocumab or placebo).
  mg/dL | 181.3 (41.89) | 216.3 (78.61) | 249.8 (86.68) | 226.0 (77.80) | 216.6 (71.84)
Non-high-density lipoprotein cholesterol (Non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] — Baseline value is defined as the last available value prior to the first dose of double-blind period (alirocumab or placebo).
  mg/dL | 124.3 (49.00) | 165.9 (75.59) | 189.4 (93.43) | 163.4 (86.88) | 159.6 (74.97)
Apolipoprotein (Apo) B100 [Mean (Standard Deviation); unit: mg/dL] — Baseline value is defined as the last available value prior to the first dose of double-blind period (alirocumab or placebo).
  mg/dL | 89.2 (27.29) | 101.0 (15.77) | 129.4 (58.27) | 103.6 (42.83) | 104.7 (37.38)
Apolipoprotein (Apo) A1 [Mean (Standard Deviation); unit: mg/dL] — Baseline value is defined as the last available value prior to the first dose of double-blind period (alirocumab or placebo).
  mg/dL | 136.3 (29.75) | 131.4 (30.02) | 154.0 (10.98) | 154.8 (20.36) | 142.7 (25.65)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Measured Serum Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 15
Description: By day 15, participants in groups A and C had received 1 subcutaneous (SC) dose of 150 mg alirocumab and participants in group B and D had received 1 SC dose of placebo. [Baseline adjusted least squares (LS) means and standard errors were obtained using analysis of covariance (ANCOVA) model specifying the treatment arm as the fixed effect and the baseline measured LDL-C value as a covariate.]
Time Frame: Baseline to Day 15
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) | PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B) | PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) | PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2: Group D)
Number analyzed (Participants) | 6 | 7 | 5 | 5
percent change | -62.48 (8.217) [lower limit 8.217] | -8.77 (7.575) [lower limit 7.575] | -48.21 (7.660) [lower limit 7.660] | -4.93 (7.660) [lower limit 7.660]
Statistical Analysis 1: Comparison: PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) vs PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B); Test type: Superiority; p = 0.0009, ANCOVA — Threshold for significance ≤ 0.05; LS Mean Difference = -53.72, 95% CI 2-sided [-79.31 to -28.12], Standard Error of Mean 11.486
Statistical Analysis 2: Comparison: PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) vs PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2: Group D); Test type: Superiority; p = 0.0056, ANCOVA — Threshold for significance ≤ 0.05; LS Mean Difference = -43.28, 95% CI 2-sided [-69.21 to 17.35], Standard Error of Mean 10.965

2. Secondary Outcome: Percent Change in Apolipoprotein (Apo) B100 From Baseline to Day 15
Description: Baseline adjusted LS means and standard errors were obtained using the same ANCOVA model as for primary endpoint specifying the treatment arm as the fixed effect and the parameter value as a covariate.
Time Frame: Baseline to Day 15
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) | PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B) | PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) | PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2: Group D)
Number analyzed (Participants) | 6 | 7 | 5 | 5
percent change | -53.33 (8.678) [lower limit 8.678] | -3.78 (8.008) [lower limit 8.008] | -47.73 (7.547) [lower limit 7.547] | -3.09 (7.547) [lower limit 7.547]
Statistical Analysis 1: Comparison: PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) vs PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B); LS means (SE), mean difference, 95% CI, and p-values were derived from ANCOVA with treatment group as factor and baseline as covariate; Test type: Superiority; p = 0.0021, ANCOVA — Threshold for significance ≤ 0.05; LS Mean Difference = -49.55, 95% CI 2-sided [-76.39 to -22.7], Standard Error of Mean 12.050
Statistical Analysis 2: Comparison: PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) vs PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2: Group D); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0045, ANCOVA — Threshold for significance ≤ 0.05; LS Mean Difference = -44.64, 95% CI 2-sided [-70.36 to 18.92], Standard Error of Mean 10.876

3. Secondary Outcome: Percent Change in Non High-Density Lipoprotein Cholesterol (Non-HDL-C) From Baseline to Day 15
Time Frame: Baseline to Day 15
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) | PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B) | PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) | PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2: Group D)
Number analyzed (Participants) | 6 | 7 | 5 | 5
percent change | -56.87 (8.217) [lower limit 8.217] | -7.50 (7.575) [lower limit 7.575] | -44.40 (7.357) [lower limit 7.357] | -4.04 (7.357) [lower limit 7.357]
Statistical Analysis 1: Comparison: PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) vs PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B); Test type: Superiority; p = 0.0016, ANCOVA — Threshold for significance ≤ 0.05; LS Mean Difference = -49.37, 95% CI 2-sided [-74.96 to -23.77], Standard Error of Mean 11.487
Statistical Analysis 2: Comparison: PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) vs PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2: Group D); Test type: Superiority; p = 0.0063, ANCOVA — Threshold for significance ≤ 0.05; LS Mean Difference = -40.36, 95% CI 2-sided [-65.12 to 15.60], Standard Error of Mean 10.471

4. Secondary Outcome: Percent Change in Total Cholesterol (Total-C) From Baseline to Day 15
Time Frame: Baseline to Day 15
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) | PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B) | PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) | PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2: Group D)
Number analyzed (Participants) | 6 | 7 | 5 | 5
percent change | -36.94 (5.203) [lower limit 5.203] | -6.18 (4.802) [lower limit 4.802] | -29.40 (4.422) [lower limit 4.422] | -7.18 (4.422) [lower limit 4.422]
Statistical Analysis 1: Comparison: PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) vs PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B); Test type: Superiority; p = 0.0017, ANCOVA — Threshold for significance ≤ 0.05; LS Mean Difference = -30.75, 95% CI 2-sided [-46.85 to -14.66], Standard Error of Mean 7.224
Statistical Analysis 2: Comparison: PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) vs PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2: Group D); Test type: Superiority; p = 0.0096, ANCOVA — Threshold for significance ≤ 0.05; LS Mean Difference = -22.23, 95% CI 2-sided [-37.11 to -7.34], Standard Error of Mean 6.294

5. Secondary Outcome: Percent Change in Apolipoprotein (Apo) B100/ ApoA-1 Ratio From Baseline to Day 15
Time Frame: Baseline to Day 15
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) | PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B) | PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) | PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2: Group D)
Number analyzed (Participants) | 6 | 7 | 5 | 5
percent change | -55.26 (7.188) [lower limit 7.188] | -5.53 (6.647) [lower limit 6.647] | -48.34 (8.090) [lower limit 8.090] | 0.99 (8.090) [lower limit 8.090]
Statistical Analysis 1: Comparison: PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) vs PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B); Test type: Superiority; p = 0.0005, ANCOVA — Threshold for significance ≤ 0.05; LS Mean Difference = -49.72, 95% CI 2-sided [-71.71 to -27.74], Standard Error of Mean 9.867
Statistical Analysis 2: Comparison: PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) vs PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2: Group D); Test type: Superiority; p = 0.0037, ANCOVA — Threshold for significance ≤ 0.05; LS Mean Difference = -49.33, 95% CI 2-sided [-76.63 to -22.03], Standard Error of Mean 11.545

ADVERSE EVENTS:
Time Frame: From the screening visit after the last alirocumab injection in the open-label period + 70 days through the end of study
Description: Observation periods for safety analyses: Pretreatment: screening to before 1st injection of alirocumab; Double-blind (DB) treatment-emergent (TE): after 1st through last in DB+70 days; Interim: after last in DB+70 days prior to 1st in open-label (OL). OL TE: after 1st through last in OL+70 days. Post: after last in OL+70 days through end of study.
Groups:
- PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2:Group D): Subjects with a GOFm in PCSK9 gene or LOFm in Apo B gene (Cohort 2: Group D) received 150 mg alirocumab SC on days 15, 29, 43, 57, and 85 and matching placebo SC on days 1, 71, and 99 during the double-blind period. Afterwards, subjects continued in an open-label extension period with 150 mg alirocumab SC twice per week (Q2W) for an additional 3 years.
- OLE Period: PCSK9 GOFm (Cohort 1) Group A & Group B: Subjects with a GOFm in PCSK9 gene (Cohort 1): alirocumab 150 mg subcutaneous (SC) injection at Week 0 (Day 1), Week 2 (Day 15), Weeks 4, 6 and 10 (matching placebo at Week 8, 12 and 14) during the double-blind period (Group A) or at Week 2 (Day 15), Weeks 4, 6, 8 and 12 (matching placebo at Week 0 [Day 1], Weeks 10 and 14) during the double-blind period (Group B). Afterwards, subjects continued in an OLE period with 150 mg alirocumab SC twice per week (Q2W) for an additional 3 years.
- OLE Period: PCSK9 GOFm/ ApoB LOFm (Cohort 2) Group C & Group D: Subjects with a GOFm in the PCSK9 gene or a LOFm in the Apo B gene (Cohort 2): alirocumab 150 mg SC injection at Week 0 (Day 1), Week 2 (Day 15), Weeks 4, 6 and 10 (matching placebo at Weeks 8, 12 and 14) during the double-blind period (Group C) or at Week 2 (Day 15), Weeks 4, 6, 8 and 12 (matching placebo at Week 0 [Day 1], 10 and 14) during the double-blind period (Group D). Afterwards, subjects continued in an OLE period with 150 mg alirocumab SC twice per week (Q2W) for an additional 3 years.
Arm/Group | PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) | PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B) | PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) | PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2:Group D) | OLE Period: PCSK9 GOFm (Cohort 1) Group A & Group B | OLE Period: PCSK9 GOFm/ ApoB LOFm (Cohort 2) Group C & Group D
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/5 | 0/5 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/7 | 0/5 | 0/5 | 3/11 | 0/10
Other Adverse Events (participants affected / at risk) | 6/6 | 6/7 | 5/5 | 4/5 | 10/11 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) (N=6) | PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B) (N=7) | PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) (N=5) | PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2:Group D) (N=5) | OLE Period: PCSK9 GOFm (Cohort 1) Group A & Group B (N=11) | OLE Period: PCSK9 GOFm/ ApoB LOFm (Cohort 2) Group C & Group D (N=10)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCSK9 GOFm: Alirocumab From Day 1 (Cohort 1: Group A) (N=6) | PCSK9 GOFm: Alirocumab From Day 15 (Cohort 1: Group B) (N=7) | PCSK9 GOFm/ApoB LOFm: Alirocumab From Day1 (Cohort 2: Group C) (N=5) | PCSK9GOFm/ApoB LOFm: Alirocumab From Day 15(Cohort 2:Group D) (N=5) | OLE Period: PCSK9 GOFm (Cohort 1) Group A & Group B (N=11) | OLE Period: PCSK9 GOFm/ ApoB LOFm (Cohort 2) Group C & Group D (N=10)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (4) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (3) | 1 (1) | 2 (4) | 1 (1) | 4 (6) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dyspesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nitrite urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peau d'orange (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.